CLINICAL TRIAL: NCT02803242
Title: COPD Patient-Powered Research Network
Acronym: COPD PPRN
Status: Recruiting | Type: Observational
Sponsor: COPD Foundation (Other)
Collaborators: Kaiser Foundation Hospitals, Center for Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: COPDPPRN
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disorder; Chronic Obstructive Lung Disease; Emphysema; Chronic Bronchitis
Keywords: copd; emphysema; bronchitis; bronchiectasis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Bronchitis; Bronchiectasis | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patient Reported Outcomes
  Other Names: Patient reported outcomes will be collected using self-report questionnaires to asses lung health status

SUMMARY:
The COPD Patient-Powered Research Network (COPD PPRN) is a patient research registry with the goal of enrolling 75,000 or more COPD patients and those at risk who are willing to share their heath information over several years and participate in research. The COPD PPRN has built an online platform to allow volunteers to enroll electronically, complete surveys, be contacted about studies they qualify for and become connected to COPD resources. The goal of the registry is to speed research to find better treatments for COPD and ultimately a cure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older that says yes to one of the following:
* COPD diagnosis
* Current or former smoker
* Family history of respiratory disease
* Symptomatic of respiratory disease

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: English speaking individuals who are over the age of 18 and have a diagnosis of COPD or fall into one of the following categories that put's them at risk - current or former smoker, environmental/occupational exposure, family history of respiratory disease or symptomatic of respiratory disease.
Sampling Method: Non-Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2014-08; Primary Completion 2025-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome Measurement Information System-29 (PROMIS-29) | 15 years
COPD Assessment Test (CAT) | 15 years
Modified Medical Research Council (MMRC) Dyspnea Scale | 15 years
Charlson Comorbidity Index (CCI) | 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- COPD Foundation, Washington D.C., District of Columbia, United States